CLINICAL TRIAL: NCT05156671
Title: Multicenter, Randomized, Double-blind, Biomarker-guided, Phase II Trial With Adrecizumab (HAM 8101) to Improve proGNosis and outcomES in Patients With Moderate to Severe COVID-19
Brief Title: Adrecizumab (HAM8101) to Improve Prognosis and Outcomes in COVID-19 Trial
Acronym: AGNES-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor recruitment.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGNES-19
Record Dates: First submitted 2021-12-02; First posted 2021-12-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Vascular Integrity; Adrecizumab; Enibarcimab; acute lung injury
MeSH Terms: conditions — COVID-19; Acute Lung Injury | interventions — enibarcimab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrecizumab (HAM 8101) (Experimental): Adrecizumab (HAM 8101) on top of standard of care. Adrecizumab (HAM8101) is a humanized IgG1 monoclonal antibody (mAb). 2 mg/kg body weight Adrecizumab diluted in up to 100 mL saline as single dose infusion.
  Interventions: Biological: Adrecizumab (HAM 8101)
- Placebo/ control substance (NaCl 0.9%) (Placebo Comparator): 100 mL saline as single dose infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Adrecizumab (HAM 8101) — Drip infusion over 60 minutes.
  Arms: Adrecizumab (HAM 8101)
Drug: Placebo — Drip infusion over 60 minutes
  Other Names: Saline
  Arms: Placebo/ control substance (NaCl 0.9%)

SUMMARY:
The clinical trial is designed as a prospective, multi-center, double-blind, randomised, placebo-controlled, interventional trial to assess safety, tolerability and efficacy of Adrecizumab (on top of SOC) in patients with COVID-19, and to evaluate if improvement of vascular integrity with Adrecizumab on top of SOC is superior to placebo/ control substance (NaCl 0.9%) on top of SOC in reduction of morbidity and mortality endpoints in patients with COVID-19.

The main reason for admission to ICU and need for mechanical ventilation of these patients is acute lung injury within a broad pneumonic spectrum, increased ventricular filling pressures and resulting congestion. It is hypothesized, that Adrenomedullin (ADM) is a key player in the (dys)-regulation of vascular integrity (Figure 2). Adrecizumab is the first-in-class humanized monoclonal anti-Adrenomedullin antibody, and acts as a long-lasting plasma Adrenomedullin enhancer stabilizing barrier function at a reasonable safety profile. The mode of action for the anti-Adrenomedullin antibody Adrecizumab has been developed on the basis of published data, own experimental data and theoretical considerations.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization with moderate to severe COVID-19, defined as fulfilling at a minimum the following clinical status category on the WHO 8-point ordinal scale: (i) "score 4" [oxygen via mask or nasal]
* Laboratory-confirmed SARS-CoV-2 infection at index hospitalisation as determined by PCR or other validated commercial or public health assay
* Bio-ADM ≥50 pg/mL or ≥30% increase until the end of the next day (with a minimum of 35 pg/mL at all)
* DPP3 ≤30 ng/mL
* Age ≥18 years at time of screening
* Body weight ≤ 150 kg at time of screening

Exclusion Criteria:

* Life expectancy less than 3 months before COVID-19 at the discretion of the Investigator
* Invasive mechanical ventilation ≥ 72 hours at time-point of randomization
* Resuscitation > 45 minutes
* Hypersensitivity to the active substance, to Adrecizumab or any of its excipients, or known serious hypersensitivity to other monoclonal antibodies
* Uncontrolled haematological/ oncological malignancies
* Pre-existing severe chronic liver disease (i.e. Child-Pugh C) before COVID-19 hospitalization
* Absolute neutropenia <500 per μL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | 90 days
  Time to clinical improvement, defined as the time from randomization to an improvement of two points (from the status at randomization) on the World Health Organisation 8-point ordinal scale or live discharge from the hospital, whichever came first.
  WHO 8-point ordinal scale
  1. Ambulatory No limitation of activities
  2. Ambulatory Limitation of activities
  3. Hospitalized, mild disease No oxygen therapy
  4. Hospitalized, mild disease Oxygen by mask or nasal cannulae
  5. Hospitalized, severe disease Non-invasive ventilation on high-flow oxygen
  6. Hospitalized, severe disease Intubation and invasive mechanical ventilation
  7. Hospitalized, severe disease Invasive mechanical ventilation and additional organ support
  8. Death -

SECONDARY OUTCOMES:
Clinical status at day 28, as measured on the WHO 8-point ordinal scale | 28 days
  Please see Outcome 1 for details on WHO 8-point ordinal scale
Survival (time-to-event) until day 28 and end of follow-up (90 days) | 90 days
Rate of invasive mechanical ventilation until day 28 and day 90 | 28 and 90 days
  defined as use of endotracheal or tracheostomy tube assisted ventilation
Length of invasive mechanical ventilation until day 28 and day 90 | 28 and 90 days
  defined as use of endotracheal or tracheostomy tube assisted ventilation
Rate of ECMO therapy until day 28 and day 90 | 28 and 90 days
Length of ECMO therapy until day 28 and day 90 | 28 and 90 days
Length of stay at ICU after application of IMP up to a total of 90 days | 90 days
Length of hospital stay after application of IMP up to a total of 90 days | 90 days
All-cause rehospitalisation within 90 days | 90 days
Rate of renal replacement therapy until day 28 and day 90 | 28 and 90 days
Change in clinical status on the WHO 8-point ordinal scale for COVID-19 at days 7, 28, and 90 | 7, 28 and 90 days
  Please see Outcome 1 for Details in WHO 8-point ordinal scale
Change in SOFA score sum (only during hospitalization on ICU) with-in 24 hours of IMP administration (start of infusion), 48 hours, day 7 post-infusion | 24 hours, 48 hours and 7 days post-infusion
Between-group difference in life quality as assessed by EQ-5D-5L at discharge, day 28, day 90 | 28 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — University Medical Center Hamburg-Eppendorf - Department of Intensive Care Medicine
Locations (13):
- Germany (13):
  - Charité, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - University Medical Center Hamburg Eppendorf, Hamburg
  - Medical School Hanover, Hanover
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar TU München, München
  - LMU München, München
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No